CLINICAL TRIAL: NCT04730531
Title: Postoperative Pain Control Using Local Wound Infiltration in Adolescent Idiopathic Surgery: A Randomized Control Trial
Brief Title: Postoperative Pain Control Using Local Wound Infiltration in Adolescent Idiopathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Craig Birch, Instructor of Orthopedic Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-P00037508
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pain; Spinal Fusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Local infiltration with 0.25% bupivacaine and epinephrine
  Interventions: Procedure: Local infiltration with 0.25% bupivacaine and epinephrine
- Control Arm (Placebo Comparator): Placebo of equal volume injectable saline
  Interventions: Procedure: Placebo of equal volume injectable saline

INTERVENTIONS:
Procedure: Local infiltration with 0.25% bupivacaine and epinephrine — The local infiltration will occur in 2 stages, separated by 30 minutes. The first dose will be injected just prior to the final tightening of set screws, decortication, and bone grafting, and will occur via multiple small volume injections 1 centimeter apart into the paraspinal musculature. The second injection will occur at an interval of 30 minutes following deep fascial closure and similarly consist of multiple small volume injections at 1 centimeter intervals into the subcutaneous tissue and skin.
  Arms: Treatment Arm
Procedure: Placebo of equal volume injectable saline — An equal volume of injectable saline will be used in the exact 2 stages as the treatment group. The first dose will be injected just prior to the final tightening of set screws, decortication, and bone grafting, and will occur via multiple small volume injections 1 centimeter apart into the paraspinal musculature. The second injection will occur at an interval of 30 minutes following deep fascial closure and similarly consist of multiple small volume injections at 1 centimeter intervals into the subcutaneous tissue and skin.
  Arms: Control Arm

SUMMARY:
Non-opioid methods of pain management following posterior spinal fusion (PSF) have become increasingly popular given the rise of opioid abuse and opioid-related deaths. Orthopedic surgery remains one of the highest prescribing subspecialties. Local wound infiltration is an effective method of acute pain management following surgical intervention and is the standard in some surgical subspecialties, however, no randomized control trials (RCT) exist in the pediatric spine literature. This would be the first (RCT) to assess the use of local would infiltration in postoperative pain control following PSF for adolescent idiopathic scoliosis patients (AIS). The primary aim of this study is to investigate the efficacy of local wound infiltration with anesthetic agents in reduction of postoperative pain scores and post-operative opioid use during hospital admission following fusion surgery in AIS patients. The proposed single-center, double-blind prospective randomized study will be conducted by recruiting patients meeting the inclusion criteria of age 10-26 years and diagnosis of AIS undergoing posterior fusion surgery. Study participants will be randomized into either a local injection of 0.25% bupivacaine with epinephrine or a placebo of equal volume injectable saline. Patient-reported outcomes will be collected at 1-, 6-, 12- and 24-months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ≥10 years old and ≤17 years old at assessment
* Diagnosis of Adolescent Idiopathic Scoliosis (AIS)
* Planned surgical treatment of progressive spinal deformity with posterior spinal fusion

Exclusion Criteria:

* Diagnosis of neuromuscular, syndromic, or congenital scoliosis
* History of known allergy to local anesthesia
* Chronic pre-operative opioid consumptions
* Any other analgesic treatment for chronic pain before surgery
* Psychiatric or neurological disorders
* Cannot fluently read or speak English

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain score | 24 hours post-operatively
  The average Visual Analog Scale pain score (on a scale of 0-100 mm) during the first 24 hours postoperatively will be computed from at most six values typically obtained every four to six hours following surgery. The higher the score, the higher the experienced pain of the individual.

SECONDARY OUTCOMES:
Average use of morphine equivalents | 24 hours post-operatively
  The average use of morphine equivalents per kilogram during the first 24 hours postoperatively. Morphine equivalents per kilogram will be also be obtained by reviewing post-anesthesia care unit reports.
Scoliosis Patient Questionnaire - Version 30 (SRS-30) | 1-, 6-, and 12-months post-operatively
  SRS-30 scores at 1-, 6-, and 12-months post-operatively. The Scoliosis Research Society (SRS-30) questionnaire is a 30-question patient reported instrument developed to evaluate health-related quality of life in patients with scoliosis. Scores from the SRS-30 are compiled into five domain scores: pain, function, self-image, mental health and satisfaction with management of scoliosis. Each domain score is reported on a scale form 1-5. The lower the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Birch, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No